CLINICAL TRIAL: NCT00470743
Title: A Randomised Controlled Trial Comparing Ibuprofen And Indomethacin For The Treatment Of The Patent Ductus Arteriosus In Very Premature Infants
Brief Title: Comparing Ibuprofen And Indomethacin For The Treatment Of The Patent Ductus Arteriosus in Very Premature Babies
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National University Hospital, Singapore (Other); Cumberland Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Quek Bin Huey, Consultant, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SQPDA02
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2009-06

CONDITIONS: Ductus Arteriosus, Patent; Very Low Birth Weight Infants
Keywords: Ibuprofen; Indomethacin; Infant, very low birth weight; Prematurity; Ductus Arteriosus, patent
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Ibuprofen; Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen (Experimental): Compare ibuprofen
  Interventions: Drug: Ibuprofen
- Normal saline (Placebo Comparator): Compared against ibuprofen -- placebo
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: Ibuprofen
  Arms: Ibuprofen
Drug: Indomethacin
  Arms: Normal saline

SUMMARY:
The purpose of the study is to determine the safety and efficacy of ibuprofen, compared with indomethacin, in the treatment for the closure of the patent ductus arteriosus in premature babies born under 29 weeks gestation

DETAILED DESCRIPTION:
According to Very Low Birth Weight (VLBW) High Risk Registration database in KKWCH, a hemodynamically significant patent ductus arteriosus (PDA) is a common problem in very premature infants born at a gestational age of 29 weeks and under, with more than 50% of them needing indomethacin treatment for closure of the PDA.

Prostaglandins play a major role in keeping the ductus patent . Indomethacin, because of its anti-prostaglandin effect via inhibition of the prostaglandin forming cyclo-oxygenase enzymes, has been used to medically close the PDA since the 1970s. Concerns with this drug relate to its effect on cerebral, renal and gastrointestinal blood flow. Necrotising enterocolitis (NEC), gastrointestinal perforation, gastrointestinal bleeding, transient or permanent renal impairment and reduced cerebral blood flow have been associated with indomethacin.

Ibuprofen treatment for PDA have been reported in the 1990s. It is as effective as indomethacin in closing the PDA. It is potentially better than indomethacin because regional blood flows were not affected. The few trials that have been done comparing intravenous ibuprofen and indomethacin involved mainly heavier very low birth weight (VLBW) infants. In a New England Journal of Medicine editorial on this subject, Clyman pointed out the need for trials involving the very immature infants to look at efficacy and safety.

The main obstacle for ibuprofen use in premature infants is the absence of a commercially available intravenous preparation. In our proposed trial a new i.v. ibuprofen preparation manufactured by Cumberland Pharmaceuticals (Nashville, Tennessee) will be used.

A Cochrane systematic review on ibuprofen for the treatment of PDA in premature infants concluded that it performed with the same effectiveness when compared to indomethacin. There was a significant decrease in the incidence of oliguria in the ibuprofen arm, with a higher risk of chronic lung disease at 28 days of life (borderline statistical significance), but not at 36 weeks.There is no biologically plausible explanation for the latter effect and this could be attributed to chance in view of this, plus the weak statistical proof. The other problem with this review was that it included trials where enteral ibuprofen was used, and this route is clearly impractical in the very premature infants which we plan to study because of the unpredictable absorption from the immature gut and their general intolerance to feeding at such an early age. The concern regarding pulmonary hypertension with the prophylactic use of ibuprofen also should not apply to our planned study where the time of administration of the drugs will be around 24 hours of age.

The potential benefits stemming from ibuprofen's biological advantage over indomethacin will be reduction in the rates of oliguria, gastrointestinal bleeding, NEC and gastrointestinal perforation. NEC and gastrointestinal perforation are conditions with serious morbidities and usually result in prolonged hospital stay and poorer neurodevelopmental outcome for the affected infants. A better drug could lead to cost savings.

Neurosensory impairment is an important outcome to monitor because indomethacin reduces cerebral blood flow. This point was also emphasized in the Cochrane systematic review mentioned above. However this will be the subject of another proposal in view of the significant additional budget needed.

The objective of the trial is to compare, the the safety and efficacy of intravenous ibuprofen treatment for the closure of the patent ductus arteriosus diagnosed via 2D echocardiography in very premature babies born under 29 weeks of gestation, with traditional therapy indomethacin.

The primary outcome measure will be the incidence of oliguria and gastric bleeding within one week after the 1st dose of treatment

ELIGIBILITY:
Inclusion Criteria:

* Infants <29 weeks gestation with a PDA diameter of >= 1.5 mm on 2Dechocardiogram
* Parental written informed consent - Parent agrees to the subject's participation in the study as indicated by parent's signature on the consent form
* Parent is willing to comply with procedures/treatment and is able to keep to scheduled study assessments

Exclusion criteria:

* Major congenital malformations in the opinion of the investigator
* Necrotising enterocolitis
* Gastrointestinal Perforation
* Systemic illness other than PDA, not fit for the trial in the opinion of the investigator
* The parent is in the opinion of the investigator, mentally or legally incapacitated
* The parent is unwilling/unable to comply to study procedures

Max Age: 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of oliguria and gastric bleeding | within one week of treatment

SECONDARY OUTCOMES:
PDA closure rates after medical treatment at time of discharge from hospital | after 1 to 2 courses of treatment
Need for repeat of the second course of medication | 48 hrs after 3rd dose of treatment
Need for surgical closure | after 1 to 2 courses of treatment
In-hospital mortality | while in-hospital
Creatinine >140umol/L within one week after the 1st dose of treatment | one week after 1st dose of treatment
Hyponatremia within one week after the 1st dose of treatment | one week after 1st dose of treatment
Gastrointestinal perforation within one week after the 1st dose of treatment | within one week after the 1st dose of treatment
Necrotising enterocolitis within one week after the 1st dose of treatment | within one week after the 1st dose of treatment
Worst grade of IVH by Day 28 of life | Day 28 of life
Pulmonary hypertension within 48hrs after 1st dose of treatment | within 48hrs after 1st dose of treatment
Chronic lung disease | Day 28 and corrected age of 36 weeks post-menstrual age
Cystic periventricular leukomalacia at day 28 of life and at term | Day 28 of life and term corrected age
Retinopathy of prematurity (Worst grade) | Within hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Quek Bin Huey, MMed MRCP, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital / National University Hospital, Singapore, Singapore